CLINICAL TRIAL: NCT05366075
Title: The Preventing Functional Decline in Acutely Hospitalized Older Patients (PREV_FUNC) Study
Acronym: PREV_FUNC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); Center for Innovative Medicine (Unknown); Konung Gustaf V:s och Drottning Victorias Frimurarestiftelse (Unknown)
Responsible Party: Principal Investigator, Anna-Karin Welmer, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FoUI-961330; 2021-01788 (Other Grant/Funding Number: FoUI-960460)
Record Dates: First submitted 2022-05-01; First posted 2022-05-09 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hospitalization; Older Adults
Keywords: Exercise; Hospitalization; Older Adults; Physical Functional Performance; Randomized Controlled Trial
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (simple exercise program) (Experimental): The intervention will include up to four sessions per day. It consists of sit-to stand exercises and walking along the corridor of the ward (for those who can walk).
  Interventions: Other: Intervention 1 (simple exercise program)
- Intervention 2 (comprehensive exercise program) (Experimental): This intervention consists of two daily sessions (morning and afternoon). The morning session includes individualized supervised progressive resistance, balance, and walking training exercises, tailored to each participant's capacity. The resistance training includes using weight cuffs, involving mainly lower-extremity muscles. Balance and gait exercises includes different exercises such as line walking, stepping practice, and walking with small obstacles. The evening session consists of functional exercises using light loads, such as knee extension and flexion, hand training with a ball, and daily walking exercises (for those who can walk).
  Interventions: Other: Intervention 2 (comprehensive exercise program)
- Control group (No Intervention): The control group will receive usual care, which may include physical rehabilitation when needed.

INTERVENTIONS:
Other: Intervention 1 (simple exercise program) — Up to four sessions per day (total duration 20-30 minutes/day). Performed at the hospital on all weekdays from baseline until hospital discharge (around 1 week). At discharge, the participants will be encouraged to continue with the exercise program at home.
  Arms: Intervention 1 (simple exercise program)
Other: Intervention 2 (comprehensive exercise program) — Two daily sessions (morning and afternoon) of 20 minutes' duration each. Performed at the hospital on all weekdays from baseline until hospital discharge (around 1 week).
  Arms: Intervention 2 (comprehensive exercise program)

SUMMARY:
This study aims to examine 1) if multicomponent exercise interventions (including both mobility and strengthening exercises) have effects on physical function compared to usual care in older adults, and 2) if a comprehensive multicomponent exercise program is more effective than a simple multicomponent exercise program including only walking and rising from a chair.

DETAILED DESCRIPTION:
This is a three-armed randomized controlled trial, with two intervention groups (comprehensive and simple exercise program) and a control group receiving usual care. Participants aged ≥75 years will be included consecutively from geriatric medical wards of hospitals in Stockholm, Sweden. Assessments will be conducted at hospital admission, discharge and three months thereafter concerning physical function (primary outcome), activities of daily living, health-related quality of life, sarcopenia, and falls. Number of re-admissions and mortality will be registered up to 1 year after discharge.

ELIGIBILITY:
Inclusion Criteria:

* ability to stand up from a sitting position independently or with minimal personal help
* ability to communicate and collaborate with the research staff

Exclusion Criteria:

* people who are not able to follow instructions
* people who by the responsible physician are assessed as not eligible to participate due to terminal illness or any major medical condition that contraindicates exercise
* those living in nursing home
* those previously included in the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Physical function | Change from baseline (hospital admission) to completion of the hospital-based exercises (at discharge around 1 week after baseline)
  Short Physical Performance Battery (Possible score: 0-12), a higher score represents a better physical function)
Physical function | Change from baseline (hospital admission) to 3 months after discharge
  Short Physical Performance Battery (Possible score: 0-12), a higher score represents a better physical function)

SECONDARY OUTCOMES:
Activities of daily living | Change from baseline (hospital admission) to completion of the hospital-based exercises (at discharge around 1 week after baseline)
  Barthel Index (Possible score: 0-100, a higher score represents a better functional ability)
Activities of daily living | Change from baseline (hospital admission) to 3 months after discharge
  Barthel Index (Possible score: 0-100, a higher score represents a better functional ability)
Health related quality of life | Change from baseline (hospital admission) to completion of the hospital-based exercises (at discharge around 1 week after baseline)
  EuroQol-5 Dimension
Health related quality of life | Change from baseline (hospital admission) to 3 months after discharge
  EuroQol-5 Dimension
Sarcopenia | Change from baseline (hospital admission) to completion of the hospital-based exercises (at discharge around 1 week after baseline)
  Defined by grip strength and calf- and arm circumferences according to the European Working Group's revised criteria on Sarcopenia in Older People
Sarcopenia | Change from baseline (hospital admission) to 3 months after discharge
  Defined by grip strength and calf- and arm circumferences according to the European Working Group's revised criteria on Sarcopenia in Older People
Number of falls | Change from baseline (hospital admission) to completion of the hospital-based exercises (at discharge around 1 week after baseline)
  According to the logbooks at the hospital
Number of falls | From hospital discharge to 3 months after discharge
  According to self-report
Mortality data | Up to 1 year after hospital discharge
  Data on vital status will be collected using administrative data
Number of readmissions | Up to 1 year after hospital discharge
  Data on readmissions will be collected using administrative data

CONTACTS AND LOCATIONS:
Locations (1):
- Anna-Karin Welmer, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandberg L, Bostrom AM, Hagstromer M, Lindgren C, Kivipelto M, Sandlund C, Welmer AK. Feasibility of the "Preventing functional decline in acutely hospitalized older patients (PREV_FUNC)" study-A three-armed randomized controlled pilot trial. PLoS One. 2024 Jun 21;19(6):e0304570. doi: 10.1371/journal.pone.0304570. eCollection 2024. PMID 38905174
- [Derived] Welmer AK, Sandberg L, Sandlund C, Bjorck C, Hagstromer M, Hamilton J, Helgstrand G, Lindgren C, Nordstrand L, Sandstedt P, Kivipelto M, Bostrom AM. Study protocol for the 'preventing functional decline in acutely hospitalised older patients (PREV_FUNC)' study: effects of two multicomponent exercise programmes on physical function - a three-armed randomised controlled trial. BMJ Open. 2023 Aug 22;13(8):e070885. doi: 10.1136/bmjopen-2022-070885. PMID 37607787